CLINICAL TRIAL: NCT00248859
Title: Determinants of Cardiac Risk Factors Modification
Brief Title: Determinants of Cardiac Risk Factor Modification in Latinos With Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Carla Boutin-Foster, MD, Study Principal Investigator, Weill Medical College of Cornell University
Other Study IDs: HL076567-01; 5K01HL076567 (NIH)
Record Dates: First submitted 2005-11-03; First posted 2005-11-04 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Depressive symptoms; Latino American
MeSH Terms: conditions — Coronary Artery Disease; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational study among Latino patients who have coronary artery disease. The goal of the study is to determine the association between having depressive symptoms and the ability to modify one's health behavior. Specifically, participate in physical activity.

DETAILED DESCRIPTION:
Specific aims: Among 213 Latino adult patients who have had coronary artery angioplasty within the past month, the specific aims of the proposed study are:

1. To determine whether patients who have more depressive symptoms at the time of angioplasty are less likely to be active in physical activity at two years. Physical activity will be measured by a survey that asks patients to describe their activities including leisure activities or housework.
2. To determine whether lower perceived social support, lower self-efficacy for engaging in physical activity, and greater perceived stress mediate the effects of depressive symptoms on participation in physical activity.

Long-term objectives: The long-term objective of this study is to use these data to develop a culturally tailored intervention to increase participation in physical activity and ultimately improve the overall health and well being of Latino adults with coronary artery disease.

Outcome: The outcome is being in the action or maintenance stage of physical activity two years after angioplasty The stage of physical activity participation will be based on the Stages of Change model. This model describes behavior change as a continuum from pre-contemplation to contemplation.

ELIGIBILITY:
Inclusion Criteria

* Patients must identify their ethnicity as Latino or Hispanic
* Patients must be able to complete a questionnaire in either English or Spanish.
* Patients must have angiographic evidence of coronary artery disease requiring angioplasty
* Patients must also be clinically stable for an interview
* Patient must be able to provide informed consent.

Exclusion criteria

* Patients who are not clinically stable such as those who had cardiac arrest, who are intubated, who have active psychosis, or who are cognitively impaired.
* Patients who are unable to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cardiovascular DiSease
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2004-08; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carla Boutin-Foster, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Joan and Sanford I. Weill Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD